CLINICAL TRIAL: NCT05369598
Title: Audiological and Quality of Life Outcomes of Anatomy Based Fitting in Patients Implanted by Robot Assisted Cochlear Implant Surgery (RACIS)
Acronym: RACIS ABF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EC-2022-022
Record Dates: First submitted 2022-03-22; First posted 2022-05-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cochlear Implants; Sensorineural Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABF fitting followed by standard fitting (Active Comparator)
  Interventions: Device: Post-operative ABF followed by fitting according to clinical standard
- Standard fitting followed by ABF fitting (Active Comparator)
  Interventions: Device: Fitting according to clinical standard followed by post-operative ABF

INTERVENTIONS:
Device: Post-operative ABF followed by fitting according to clinical standard — Cochlear implant will be fitted first with anatomy-based fitting for 6 months and followed by default fitting for 2 months.
  Arms: ABF fitting followed by standard fitting
Device: Fitting according to clinical standard followed by post-operative ABF — Cochlear implant will be fitted first with default fitting for 6 months and followed by anatomy-based fitting for 2 months.
  Arms: Standard fitting followed by ABF fitting

SUMMARY:
Severe to profound hearing loss affects 0,8% of the global population. For these people, a conventional hearing aid often does not provide sufficient benefit. However, these people can benefit from a cochlear implant (CI). A CI needs to be individually programmed (fitted) for each recipient. A fitting "map" is defined as a set of electrical parameters that are individually adapted to a recipient's needs to achieve optimal sound perception. At present, most CI recipients are fitted with a default frequency allocation map that doesn't take individual variability in size and shape of the cochlea into account. In this study, a fitting strategy based on the post-operative CT scan, that will allow the audiologist to set a frequency-band distribution for CI fitting that may be more closely aligned to the natural tonotopic frequency distribution of a normal hearing cochlea, will be evaluated. This study will focus on patients that are already implanted with the HEARO robotic system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Post-lingual onset of severe to profound sensory-neural hearing loss in the implanted ear(s)
* Subject implanted by Robot Assisted Cochlear Implant Surgery (RACIS)
* Subject implanted with MED-EL cochlear implant(s) with Flex28, Flex 26 or FlexSoft electrode to obtain maximum cochlear coverage
* Subject planned to receive a MED-EL SONNET 2 or RONDO 3 audio processor on the newly implanted side
* Subject is either a user with unilateral implantation, bilateral implantation or a bimodal CI user (unilateral CI user with contralateral ear adequately fitted with a hearing aid)
* Pre- operative and post-operative CT scan of the temporal bone available
* Pre-operative result of pure-tone audiometry, speech test in quiet and in noise available
* Audio processor not yet activated on the newly implanted side
* Minimum of 10 active channels can be activated
* Fluent in the language of the test centre (Dutch or French)
* Signed and dated ICF before the start of any study-specific procedure

Exclusion Criteria:

* Subject is a Single-Sided Deafness (SSD) CI user
* Subject is an Electric Acoustic Stimulation (EAS) user (with an EAS audio processor)
* Lack of compliance with any inclusion criteria
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Speech recognition in noise: Speech Reception Threshold (SRT) in dB SNR | 3 months post- activation
Speech recognition in noise: Speech Reception Threshold (SRT) in dB SNR | 6 months post- activation
Speech recognition in noise: Speech Reception Threshold (SRT) in dB SNR | 8 months post-activation

SECONDARY OUTCOMES:
Speech recognition in quiet: Percentage correctly identified phonemes | 3 months post-activation
Speech recognition in quiet: Percentage correctly identified phonemes | 6 months post-activation
Speech recognition in quiet: Percentage correctly identified phonemes | 8 months post-activation
Speech discrimination: Number of correctly discriminated pairs of phonemes | 3 months post- activation
Speech discrimination: Number of correctly discriminated pairs of phonemes | 6 months post- activation
Speech discrimination: Number of correctly discriminated pairs of phonemes | 8 months post- activation
Pure-tone audiometry with CI: Hearing thresholds between 125Hz and 8 kHz (dB HL) | 1 month post- activation
Pure-tone audiometry with CI: Hearing thresholds between 125Hz and 8 kHz (dB HL) | 3 month post- activation
Pure-tone audiometry with CI: Hearing thresholds between 125Hz and 8 kHz (dB HL) | 6 months post- activation
Pure-tone audiometry with CI: Hearing thresholds between 125Hz and 8 kHz (dB HL) | 8 months post- activation
Patient reported outcome- Nijmegen Cochlear Implant Questionnaire (NCIQ): Total score and score in the physical, psychological and social domain | Baseline at activation
  The physical domain comprises three subdomains, namely Basic sound perception, Advanced sound perception, and Speech production. The Psychological domain contains the subdomain Self-esteem and the Social domain handles questions about Activity limitations and Social interactions. Each subdomain covers 10 statements. Each statement is rated on a 5-point Likert scale ranging from "Never" to "Always" (Statement 1-55) or from "No" to "Quite well" (Statement 56-60). Scores for the subdomains will be computed by transforming the answer categories (1-5) for all items: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100 and by adding together the 10-item scores of each subdomain and dividing by the number of completed items.For each subdomain, the score ranges between 0-100 and a higher score indicates a better outcome.
Patient reported outcome- Nijmegen Cochlear Implant Questionnaire (NCIQ): Total score and score in the physical, psychological and social domain | 3 months post- activation
  The physical domain comprises three subdomains, namely Basic sound perception, Advanced sound perception, and Speech production. The Psychological domain contains the subdomain Self-esteem and the Social domain handles questions about Activity limitations and Social interactions. Each subdomain covers 10 statements. Each statement is rated on a 5-point Likert scale ranging from "Never" to "Always" (Statement 1-55) or from "No" to "Quite well" (Statement 56-60). Scores for the subdomains will be computed by transforming the answer categories (1-5) for all items: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100 and by adding together the 10-item scores of each subdomain and dividing by the number of completed items.For each subdomain, the score ranges between 0-100 and a higher score indicates a better outcome.
Patient reported outcome- Nijmegen Cochlear Implant Questionnaire (NCIQ): Total score and score in the physical, psychological and social domain | 6 months post- activation
  The physical domain comprises three subdomains, namely Basic sound perception, Advanced sound perception, and Speech production. The Psychological domain contains the subdomain Self-esteem and the Social domain handles questions about Activity limitations and Social interactions. Each subdomain covers 10 statements. Each statement is rated on a 5-point Likert scale ranging from "Never" to "Always" (Statement 1-55) or from "No" to "Quite well" (Statement 56-60). Scores for the subdomains will be computed by transforming the answer categories (1-5) for all items: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100 and by adding together the 10-item scores of each subdomain and dividing by the number of completed items.For each subdomain, the score ranges between 0-100 and a higher score indicates a better outcome.
Patient reported outcome: Nijmegen Cochlear Implant Questionnaire (NCIQ): Total score and score in the physical, psychological and social domain | 8 months post- activation
  The physical domain comprises three subdomains, namely Basic sound perception, Advanced sound perception, and Speech production. The Psychological domain contains the subdomain Self-esteem and the Social domain handles questions about Activity limitations and Social interactions. Each subdomain covers 10 statements. Each statement is rated on a 5-point Likert scale ranging from "Never" to "Always" (Statement 1-55) or from "No" to "Quite well" (Statement 56-60). Scores for the subdomains will be computed by transforming the answer categories (1-5) for all items: 1 = 0, 2 = 25, 3 = 50, 4 = 75, and 5 = 100 and by adding together the 10-item scores of each subdomain and dividing by the number of completed items. For each subdomain, the score ranges between 0-100 and a higher score indicates a better outcome.
Patient reported outcome- Speech, Spatial and Qualities of Hearing scale (SSQ12): Total score and score in the speech, spatial and quality domain | Baseline at activation
  The 12 items of this questionnaire are rated on a visual analog scale from 0 to 10 and the overall score is calculated by taking the average of the scores on these 12 items.For the overall score and the score on each subdomain, the score ranges between 0-10 and a higher score indicates a better outcome.
Patient reported outcome- Speech, Spatial and Qualities of Hearing scale (SSQ12): Total score and score in the speech, spatial and quality domain | 3 months post- activation
  The 12 items of this questionnaire are rated on a visual analog scale from 0 to 10 and the overall score is calculated by taking the average of the scores on these 12 items.For the overall score and the score on each subdomain, the score ranges between 0-10 and a higher score indicates a better outcome.
Patient reported outcome- Speech, Spatial and Qualities of Hearing scale (SSQ12): Total score and score in the speech, spatial and quality domain | 6 months post- activation
  The 12 items of this questionnaire are rated on a visual analog scale from 0 to 10 and the overall score is calculated by taking the average of the scores on these 12 items.For the overall score and the score on each subdomain, the score ranges between 0-10 and a higher score indicates a better outcome.
Patient reported outcome- Speech, Spatial and Qualities of Hearing scale (SSQ12): Total score and score in the speech, spatial and quality domain | 8 months post- activation
  The 12 items of this questionnaire are rated on a visual analog scale from 0 to 10 and the overall score is calculated by taking the average of the scores on these 12 items.For the overall score and the score on each subdomain, the score ranges between 0-10 and a higher score indicates a better outcome.
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | Baseline at activation
  The 19 items are rated on a 7-point Likert scale ranging from always (99%) to never (1%). To calculate the overall score the corresponding numerical value of each item (from always = 7 to never = 1) is added. Uncompleted items and the response option "not applicable" correspond to 0 in this calculation. A total score of less than 30, 30-59, 60-89, 90-109, and 110-133 is respectively classified as a very poor, poor, moderate, good, and very good self-perceived auditory benefit.
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 3 months post- activation
  The 19 items are rated on a 7-point Likert scale ranging from always (99%) to never (1%). To calculate the overall score the corresponding numerical value of each item (from always = 7 to never = 1) is added. Uncompleted items and the response option "not applicable" correspond to 0 in this calculation. A total score of less than 30, 30-59, 60-89, 90-109, and 110-133 is respectively classified as a very poor, poor, moderate, good, and very good self-perceived auditory benefit.
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 6 months post- activation
  The 19 items are rated on a 7-point Likert scale ranging from always (99%) to never (1%). To calculate the overall score the corresponding numerical value of each item (from always = 7 to never = 1) is added. Uncompleted items and the response option "not applicable" correspond to 0 in this calculation. A total score of less than 30, 30-59, 60-89, 90-109, and 110-133 is respectively classified as a very poor, poor, moderate, good, and very good self-perceived auditory benefit.
Patient reported outcome- Hearing Implant Sound Quality Index (HISQUI): Total score and classification of self-perceived auditory benefit | 8 months post- activation
  The 19 items are rated on a 7-point Likert scale ranging from always (99%) to never (1%). To calculate the overall score the corresponding numerical value of each item (from always = 7 to never = 1) is added. Uncompleted items and the response option "not applicable" correspond to 0 in this calculation. A total score of less than 30, 30-59, 60-89, 90-109, and 110-133 is respectively classified as a very poor, poor, moderate, good, and very good self-perceived auditory benefit.

OTHER OUTCOMES:
Evaluation of electrode contact location: Degrees of deviation | 8th months post activation

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Topsakal, Prof., Principal Investigator — UZB-VUB
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No